CLINICAL TRIAL: NCT06160778
Title: Intravenous Ketorolac Vs. Morphine In Children Presenting With Acute Abdominal Pain And/or Suspected Appendicitis: A Multi-centre Non-Inferiority Randomized Controlled Trial
Brief Title: Intravenous Ketorolac Vs. Morphine In Children With Acute Abdominal Pain
Acronym: KETOAPP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-0952
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2023-11

CONDITIONS: Acute Pain; Abdomen, Acute; Abdominal Pain; Appendicitis; Emergencies; Child, Only
MeSH Terms: conditions — Acute Pain; Abdomen, Acute; Abdominal Pain; Appendicitis; Emergencies | interventions — Ketorolac Tromethamine; Morphine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Two parallel interventional groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double dummy design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketorolac Tromethamine (Experimental): Ketorolac tromethamine, an NSAID belonging to a group of non-opioid analgesics that inhibit the synthesis of prostaglandins and thromboxanes with strong analgesic and anti-inflammatory properties. It is the only non-opioid parenteral non-sedating analgesic available in Canada for use to treat acute pain in the emergency department.
  Interventions: Drug: Ketorolac Tromethamine; Drug: normal saline
- Morphine Sulfate (Active Comparator): An intravenous opioid that is commonly used as part of usual care for treament of pain in patients with acute abdominal pain and suspected appendicitis.
  Interventions: Drug: Morphine Sulfate; Drug: Normal saline

INTERVENTIONS:
Drug: Ketorolac Tromethamine — Intravenous ketorolac given at 0.5 mg/kg of body weight up to a maximum of 30 mg in a single dose.
  Arms: Ketorolac Tromethamine
Drug: Morphine Sulfate — Intravenous morphine given at 0.1 mg/kg of body weight up to a maximum of 5 mg in a single dose.
  Arms: Morphine Sulfate
Drug: normal saline — Intravenous normal saline placebo (labelled as morphine) given at 0.1 mg/kg of body weight up to a maximum of 5 mg in a single dose.
  Other Names: Morphine Sulfate Placebo
  Arms: Ketorolac Tromethamine
Drug: Normal saline — Intravenous normal saline placebo (labelled as ketorolac) given at 0.5 mg/kg of body weight up to a maximum of 30 mg in a single dose.
  Other Names: Ketorolac Tromethamine Placebo
  Arms: Morphine Sulfate

SUMMARY:
Appendicitis is a common condition in children 6-17 years of age, and the top reason for emergency surgery in Canada. Children with appendicitis can have very bad pain in their belly. Children often need pain medications given to them through a needle in their arm called an intravenous (IV). The most common IV pain medication is a type of opioid called morphine. We know that opioids work well to improve pain, but there are risks and side effects when taking them. There are non-opioid medications that doctors can give to patients, like ketorolac. Ketorolac helps decrease inflammation and pain and has fewer side effects when a patient takes it for a short period of time. Our past and present overuse of opioids, driven by an unproven assumption that opioids work best for pain, resulted in an Opioid Crisis and doctors are now looking for alternatives. To do this, we need to prove that there are other options to treat children's pain that are just as good as opioids, with less side effects.

The goal of our study is to discover if school aged children who arrive at the emergency department with belly pain, improve just as much with ketorolac as they do with morphine. To answer this question, we will need a very large number of patients in a study that includes several hospitals across Canada. With a flip of a coin, each participant will either get a single dose of morphine or a single dose of ketorolac. To make sure that our pain assessment is impartial, no one will know which medicine the child received except the pharmacist who prepared the medicine.

DETAILED DESCRIPTION:
Background: Appendicitis, the most common surgical diagnosis in Canadian children aged 6-17 years, accounts for ~8000 admissions annually. Despite an ongoing opioid crisis, prescription narcotics remain a mainstay analgesic for children with suspected appendicitis. Ketorolac, a non-steroidal anti-inflammatory drug (NSAID), which has a safer adverse event (AE) profile than opioids, is commonly used in emergency departments (EDs) for adults; however, use in children is considered off label due to a lack of randomized trials in this patient population. We propose a multi-centre clinical trial to address this knowledge gap,informed by our team's successful pilot trial.

Specific Aim 1: To determine if administering intravenous (IV) ketorolac is non inferior to IV morphine in reducing mean pain scores in children with suspected appendicitis.

Hypothesis: IV ketorolac will be non-inferior to IV morphine

Specific Aim 2: To determine between group differences in rates of AEs. Hypothesis: IV ketorolac will be associated with less AEs than IV morphine.

Design: A randomized quadruple blind (participant, clinician, outcome assessor, investigator) parallel group double-dummy trial in 4 Canadian pediatric EDs. Eligible patients will be 6-17 years with 5-days of moderate-severe pain (vNRS ≥5 ) being investigated for suspected appendicitis, with intravenous (IV) access, will be randomized to either:

1. IV ketorolac 0.5 mg/kg up to 30 mg (intervention) + IV morphine placebo (normal saline), or
2. IV morphine 0.1 mg/kg up to 5 mg (active control) + IV ketorolac placebo (normal saline).

Primary outcome: Between-group mean difference in pain on the vNRS at 60 minutes following administration.

Safety outcome: Proportion of children experiencing AEs related to study drug administration.

Secondary Outcomes: Between-group differences: (1) pain relief as measured on vNRS at 30, 90 and 120 minutes and at 6-8 hours; (2) proportion who achieves a 2-point vNRS (minimal important difference) pain score reduction at 60 and 120 minutes; (3) proportion of patients who change their baseline pain category (vNRS: mild 0-3, moderate 4-6, severe ≥7) at each time point; (4) time to effective analgesia as measured by the time when vNRS of <3 is achieved (5) proportion of patients requiring additional analgesia; (6) total opioids administered (i.e., morphine equivalent mg/kg within 8 hours of treatment); (7) frequency of specific types of AEs (e.g., dizziness); (8) frequency of delayed appendicitis diagnosis; and (9) Ramsay Sedation Score at 30, 60, 90 and 120 minutes.

Sample size:With a non-inferiority margin of 1.0 (50% of the minimal important difference), 600 participants would give a power of 0.9 (1- β) to establish non-inferiority of ketorolac vs. morphine (significance level α = 0.05).

ELIGIBILITY:
Inclusion Criteria:

1. Age 6 to 17 years
2. Abdominal pain ≤5 days duration
3. Acute abdominal pain that is being investigated (suspected) by the clinical team for appendicitis
4. Patient with IV cannula in situ or ordered
5. Currently experiencing moderate to severe abdominal pain at rest or with movement: self-reported pain score ≥5 using the verbal Numerical Rating Scale

Exclusion Criteria:

1. Previous enrollment in the trial
2. NSAID use within 3 hours and/or opioid use within 1 to 2 hours (1 hour post-IV or intra-nasal fentanyl and 2 hours post IV morphine).
3. Children who need immediate resuscitation, are hemodynamically unstable as deemed by the clinical team or have a Canadian Triage Assessment Score of 1
4. Significant caregiver and/or child cognitive impairment precluding the ability to complete study questions.
5. Chronic pain requiring daily analgesic use: confounding as response to analgesics maybe altered.
6. History of severe undiagnosed gastrointestinal bleeding requiring medical intervention, peptic or duodenal ulcer disease or inflammatory bowel disease, coagulation disorders, prior cerebrovascular bleeding, known arterio-vascular malformations. History of minor gastrointestinal bleeding from conditions such as resolved fissures, polyps or allergic colitis will not exclude patients from participating.
7. History of chronic and active interstitial kidney disease
8. History of chronic and active hepatocellular disease: ketorolac is metabolized by the liver.
9. Known or suspected pregnancy at the time of enrollment or breastfeeding females
10. Known hypersensitivity to NSAIDs or opioids.
11. Absence of a parent/guardian for children who are <16 years of age if they are not a mature minor.
12. Inability to obtain consent due to a language barrier and the absence of language translator in person or by a phone translation service available in the ED.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 495 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Pain relief as measured on the verbal numerical rating scale | 60 minutes post drug administration
  Between group mean differences in pain as measured on an 11-point verbal Numerical Rating Scale (0 is no pain and 10 is worst pain ever)

SECONDARY OUTCOMES:
Pain relief as measured on the verbal numerical rating scale | 30 minutes post drug administration
  Between group mean differences in pain as measured on an 11-point verbal
Pain relief as measured on the verbal numerical rating scale | 90 minutes post drug administration
  Between group mean differences in pain as measured on an 11-point verbal
Pain relief as measured on the verbal numerical rating scale | 120 minutes post drug administration
  Between group mean differences in pain as measured on an 11-point verbal
Pain relief as measured on the verbal numerical rating scale | 6 hours post drug administration
  Between group mean differences in pain as measured on an 11-point verbal
Pain relief as measured on the verbal numerical rating scale during the ultrasound diagnostic | up to 6 hours post drug administration
  score from 0-10 on verbal numerical rating scale
Proportion who achieve the minimal important difference for pain relief | 60 minutes post drug administration
  Proportion of participants who achieves the 2-point verbal Numerical Rating Scale minimal important difference pain score reduction
Proportion who achieve the minimal important difference for pain relief | 120 minutes post drug administration
  Proportion of participants who achieves the 2-point verbal Numerical Rating Scale minimal important difference pain score reduction
Change in baseline pain category | 30 minutes post drug administration
  Proportion of participants who change the severity of their baseline pain category. Pain categories on the verbal numerical rating scale as follows: mild = 0 to 4, moderate = 5 to 7, severe >7)
Change in baseline pain category | 60 minutes post drug administration
  Proportion of participants who change the severity of their baseline pain category. Pain categories on the verbal numerical rating scale as follows: mild = 0 to 4, moderate = 5 to 7, severe >7)
Change in baseline pain category | 90 minutes post drug administration
  Proportion of participants who change the severity of their baseline pain category. Pain categories on the verbal numerical rating scale as follows: mild = 0 to 4, moderate = 5 to 7, severe >7)
Change in baseline pain category | 120 minutes post drug administration
  Proportion of participants who change the severity of their baseline pain category. Pain categories on the verbal numerical rating scale as follows: mild = 0 to 4, moderate = 5 to 7, severe >7)
Change in baseline pain category | 6 hours post drug administration
  Proportion of participants who change the severity of their baseline pain category. Pain categories on the verbal numerical rating scale as follows: mild = 0 to 4, moderate = 5 to 7, severe >7)
Time to effective analgesia | up to 6 hours post drug administration
  Duration of time from time of drug administration to time at which a verbal Numerical Rating Scale ≤3 is achieved.
Additional analgesia requirment | up to 6 hours post drug administration
  Proportion of participants requiring any additional analgesia in each trial arm
Total opioids administered | up to 8 hours post drug administration
  total morphine-equivalent mg/kg administered for all trial participants
Ramsay sedation score | 30 minutes post drug administration
  Assessment of sedation levels post drug administration; score is 1-6 (1 is alert, 6 is not responsive)
Ramsay sedation score | 60 minutes post drug administration
  Assessment of sedation levels post drug administration; score is 1-6 (1 is alert, 6 is not responsive)
Ramsay sedation score | 90 minutes post drug administration
  Assessment of sedation levels post drug administration; score is 1-6 (1 is alert, 6 is not responsive)
Ramsay sedation score | 120 minutes post drug administration
  Assessment of sedation levels post drug administration; score is 1-6 (1 is alert, 6 is not responsive)
Adverse events per participant | up to 6 hours post drug administration
  Frequency of specific adverse event occurrence per participant enrolled
Frequency of each specific adverse event | up to 6 hours post drug administration
  Frequency of each specific adverse event occurrence

OTHER OUTCOMES:
Appendix visualization on ultrasound | post-randomization and up to 8 hours post-intervention.
  proportion of participants who had the appendix visualized on ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Eltorki, MBChB, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital Emergency Department, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
At the completion of the study and publication of main manuscript, anonymized participant data can be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: within 10 years of study completion